CLINICAL TRIAL: NCT03990194
Title: Real-life Observational Study of Patients After 3-months of Leuprorelin 5mg Implant and Evaluation of Coping Strategies Among Patients With Prostate Cancer: LEPTO STUDY
Brief Title: Real-life Study of Patients After 3-months of Leuprorelin 5mg Implant in Prostate Cancer
Acronym: LEPTO
Status: Withdrawn | Type: Observational
Why Stopped: Internal decision
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Other Study IDs: Leptoprol- FR-NIS 0023
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Leuprolide Acetate — Administration of Leptoprol implant every 3 months
  Other Names: Leptoprol 5 mg

SUMMARY:
To improve the management of patients suffering from prostate cancer, Laboratoires BOUCHARA-RECORDATI wish to set up an observational study to document, in daily practice, and over a large population, the profile and clinical and biological follow-up of patients undergoing leuprorelin 5 mg implant as well as the conditions for implant placement. The evolution of these prostate cancer patients will be monitored on the basis of data available in daily practice, including testosterone values, PSA values, and factors that may influence disease progression, in order to objectify whether the observed results are consistent with those described in the clinical studies.

DETAILED DESCRIPTION:
To improve the management of patients suffering from prostate cancer, Laboratoires BOUCHARA-RECORDATI wish to set up an observational study to document, in daily practice, and over a large population, the profile and clinical and biological follow-up of patients undergoing leuprorelin 5 mg implant as well as the conditions for implant placement. The evolution of these prostate cancer patients will be monitored on the basis of data available in daily practice, including testosterone values, PSA values, and factors that may influence disease progression, in order to objectify whether the observed results are consistent with those described in the clinical studies.

The psychological dimension of the management of patients with prostate cancer will also be addressed by evaluating the strategies used by patients to cope with their prostate cancer [(Prostate Cancer Patients' Coping Strategies Questionnaire (PCPCSQ)].

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate cancer for whom the physician has decided to prescribe hormone therapy by subcutaneous leuprorelin implant 5 mg (Leptoprol®).

Exclusion Criteria:

* Patient who have already participated in another study or those who do not wish to participate in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer for whom the physician has decided to prescribe hormone therapy by subcutaneous leuprorelin implant 5 mg (Leptoprol®).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
The percentage of prostate cancer patients at 3 months who attained a testosteronemia threshold of ≤ 0.5 ng/mL following a 3-month treatment with leuprorelin 5 mg implant | 3 months
  The percentage of prostate cancer patients who attained a testosteronemia threshold of ≤ 0.5 ng/mL following a 3-month treatment with leuprorelin 5 mg implant will be evaluated at 3 months and at 6 months of follow-up

IPD SHARING:
Plan to Share IPD: No